CLINICAL TRIAL: NCT05459207
Title: Association Among Body Composition, Chronic Pain, Evoked Pain Sensitivity, and Adiposity-related Systemic Inflammation in Individuals With Spinal Cord Injury
Brief Title: Association Between Body Composition and Pain in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Elizabeth Felix, Research Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20211078; 90SCIMS0013 (Other Grant/Funding Number: National Institute for Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pain; Inflammatory Response
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Fat Meal, Followed by High Fat Meal Group (Experimental): Participants will receive a moderate fat meal, followed by a high fat meal approximately seven days apart.
  Interventions: Other: Moderate Fat Meal; Other: High Fat Meal
- High Fat Meal, Followed by Moderate Fat Meal Group (Experimental): Participants will receive a high fat meal, followed by a moderate fat meal approximately seven days apart.
  Interventions: Other: Moderate Fat Meal; Other: High Fat Meal

INTERVENTIONS:
Other: Moderate Fat Meal — A liquid meal consisting of powdered protein and complex carbohydrates blended with coconut oil and peanut butter in ratios required to achieve the desired calorie and macronutrient distributions of a normal/moderate fat meal.
Other: High Fat Meal — A liquid meal consisting of powdered protein and complex carbohydrates blended with coconut oil and peanut butter in ratios required to achieve the desired calorie and macronutrient distributions of a high-fat meal.

SUMMARY:
The purposes of the study are to quantify and compare relationships among acute changes in inflammatory markers and evoked pain sensitivity after a high-fat meal (HFM) challenge, compared to a moderate-fat meal challenge, and explore the influence of body composition on these responses, in individuals with chronic spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* SCI occurring at least 2 years prior to study entry
* Neurological level of injury (LOI) between C4 and L2
* American Spinal Injury Association Impairment Scale (AIS) A-D
* English-speaking.

Exclusion Criteria:

* Cognitive dysfunction that limits ability to adequately understand the risks of the study or are otherwise unable to consent
* Health conditions associated with chronic systemic inflammation unrelated to weight or adiposity (e.g., systemic autoimmune diseases, recurrent or active urinary tract infection, pressure injury > Stage 2)
* Conditions that preclude measurement of body composition by dual-energy x-ray absorptiometry (DXA; e.g., lower limb contracture > 15 degrees)
* Inability to obtain free-flowing blood from a superficial forearm or hand vein
* Pregnant women
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
peak change in Interleukin (IL)-6 | at 0, 40, 80, 160, 240, 320, and 400 minutes post meal ingestion
  analysis of blood samples taken after ingestion of meal challenge for level of IL-6 in picograms/milliliter
peak change in evoked pain sensitivity | at 0, 40, 80, 160, 240, 320, and 400 minutes post meal ingestion
  measures of heat pain threshold (degrees Celcius), using the ascending method of limits via a 30mm2 surface thermode, obtained after ingestion of meal challenge

SECONDARY OUTCOMES:
correlation coefficient between changes in IL-6 and evoked pain sensitivity | at 0, 40, 80, 160, 240, 320, and 400 minutes post meal ingestion
  correlation coefficient for relationship between changes in IL-6 and heat pain thresholds across time

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Felix, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No